CLINICAL TRIAL: NCT02016599
Title: Delineating the Effects of Transitional Circulation Physiology on Extremely Low Birth Weight (ELBW) Infants
Brief Title: Effects of Transitional Circulation in ELBW Infants
Status: Active, not recruiting | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Danielle R Rios, Professor, University of Iowa
Other Study IDs: 201911158; 1K23HL130522-01 (NIH)
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Neonatal Prematurity; Hypotension
Keywords: Hypotension; Low blood pressure; Neonate; Extremely Low Birth Weight Infant
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken to assess the lactate, troponin, and creatinine levels. These samples will be destroyed once analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Initial cohort: Initial cohort used to develop a series of multivariate clinical deterioration indices using monitoring modalities and biospecimen collection
  Interventions: Other: Monitoring and biospecimen collection
- Validation cohort: Separate cohort of infants used to validate the clinical deterioration indices using monitoring modalities and biospecimen collection
  Interventions: Other: Monitoring and biospecimen collection

INTERVENTIONS:
Other: Monitoring and biospecimen collection — The study team will use monitoring methods normally used in the NICU (physical exams, echocardiograms, and ECG) and some new monitoring methods (Near-infrared spectroscopy or NIRS) to find out all the changes that a baby's heart and lungs go through during the first week after delivery. In addition, blood samples will be taken to assess lactate, troponin, and creatinine levels.

SUMMARY:
Prematurity is a very important problem in this country. Prematurity can cause problems with organ (such as the brain, heart, kidneys) growth and development. A very important part of keeping premature babies healthy is ensuring good blood flow to all of these organs.

Some premature babies have problems with their hearts and getting enough blood out to the rest of their bodies. This problem is referred to as hypotension (low blood pressure) and is found by looking at blood test values and while examining the baby. These babies will need medications to help their heart deliver blood to all of the important areas in their bodies.

Babies who have hypotension requiring medications tend to have more problems than premature babies that don't need hypotension medication. Some of these problems include a higher risk of bleeding into their brain, kidney problems, liver problems, intestinal (gut) problems causing difficulty tolerating feeds, and a very dangerous infection of their intestines. Some long term effects include hearing loss, developmental delay, and learning problems in the future that are worse than other premature babies who did not have hypotension. Hypotensive premature babies also have a higher risk of death.

The cause of hypotension in the first week of life is still not known. We know that babies have to get used to being in the outside world instead of in the womb. A lot of changes with the heart and lungs have to happen for them to not be affected by that transition. If we could gain a better understanding of those changes, we might be able to prevent some of these issues from happening.

This study will look closely at premature babies with and without hypotension to assess the heart and lung changes in the first week of life. To do this, we will use monitoring machines and tests to get a better idea of all the changes that happen. This information will help all neonatologists who care for premature babies.

DETAILED DESCRIPTION:
Screening Phase: The subject's parents/guardians/legally authorized representative will be approached if the infant's birth weight makes them eligible for this research study.

Study Phase: During this study, we will use the monitoring methods normally used in the Neonatal Intensive Care Unit (NICU) and some new monitoring methods to find out all the changes that the infant's heart and lungs go through during the first week after delivery. During this period the study doctor and staff will:

1. Collect demographic (age, race, ethnicity) and labor/delivery information.
2. Perform serial physical exams to evaluate the infant's skin.
3. Take several blood samples (2-3 drops per sample) to measure the lactate, troponin, and creatinine levels. These blood samples will be taken 1-4 times a day.
4. Perform Echocardiograms (ultrasound of the heart) on a daily or more or less frequent basis. In between echocardiograms, we will monitor cardiac output with a non-invasive monitor using leads similar to those used for regular heart rate monitoring in the NICU. These tests are being done solely for research purposes and will be paid for by the study.
5. Measure the amount of blood flow reaching the infant's brain and kidneys using a near-infrared spectroscopy (NIRS) machine. This test is being done solely for research purposes and will be paid for by the study.
6. Perform Electrocardiograms (ECGs) to monitor how much blood flow is reaching the infant's heart. The sticky pads required for this test will be attached to the infant's chest as part of his/her routine care. For the purposes of this study, we will continuously monitor the machine to record the results.
7. Measure the amount of blood flowing in one of the arteries in the brain using cerebral Doppler ultrasound
8. Record results from any other monitoring tools the infant's doctor is using as part of his/her routine care. This will help us identify patterns that might lead to issues in premature babies. We will also be studying the effects of any medications the infant's doctor prescribes; especially those used for low blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Infant born at less than or equal to 1000 grams
* Admitted to NICU

Exclusion Criteria:

* Infant does not meet inclusion criteria
* Infant has life-threatening congenital defect
* Infant has congenital hydrops

Max Age: 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All ELBW infants are eligible for enrollment. There will not be a placebo group. Data from the first 100 patients will be used to develop the clinical deterioration indices and data from the next 100 patients will be used to validate the indices.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-09-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Quantify physiologic changes during transitional circulation | 7 days
  Develop a series of multivariate clinical deterioration indices which can be evaluated in real-time to provide continuous and calibrated measurements of likelihood of experiencing an outcome

SECONDARY OUTCOMES:
Quantify cardiac output | 7 days
  Quantify cardiac output during normal transitional circulation
Quantify the differences in perfusion of end organs | 7 days
  Quantify the differences in perfusion of end organs during transitional circulation
Measure cardiopulmonary interaction patterns | 1 year
  Measure cardiopulmonary interaction patterns during the transitional circulation and periods of hemodynamic instability to serve as forewarning of impending crisis
Quantify the change in degree of systemic perfusion | 7 days
  Quantify the change in the degree of systemic perfusion prior to and after vasoactive medication usage.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle R Rios, MD, MS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No